CLINICAL TRIAL: NCT05513521
Title: Velocity- Versus Load-based Training on Muscle Quality and Performance in Older Persons
Brief Title: Speed-specific Training and Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220489
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-08

CONDITIONS: High-Intensity Interval Training; Resistance Training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Compare velocity-based interval resistance training to load-based resistance training
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know intervention group membership.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-velocity interval training (Experimental): Subjects will be provided high-speed, low-load training to target improvements in velocity.
  Interventions: Other: High-velocity interval training
- Resistance training (Experimental): Subjects will be provided low-speed, high-load training to target improvements in velocity
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: High-velocity interval training — For the velocity training protocol, the 11 exercises will be completed at 40% of their 1RM. In the first three weeks of training, the loading volume will be increased gradually. During week one participants will complete one set of each exercise. Week two will consist of two sets, and weeks 3-12, three sets. Keiser pneumatic resistance machines are interfaced with a laboratory computer, which allows the transfer and analysis of data including force, velocity, and power.
  Arms: High-velocity interval training
Other: Resistance training — For the load training protocol, the 11 exercises will be completed at 79% of their 1RM. In the first three weeks of training, the loading volume will be increased gradually. During week one participants will complete one set of each exercise. Week two will consist of two sets, and weeks 3-12, three sets. Keiser pneumatic resistance machines are interfaced with a laboratory computer, which allows the transfer and analysis of data including force, velocity, and power.
  Arms: Resistance training

SUMMARY:
The investigators propose to compare the effects of a 12-week load resistance training program to a velocity resistance training program on ultrasound measures of quadriceps muscle quality in a healthy, older adult population. As secondary measures, The investigators propose to compare the effects of these exercise programs on maximal strength, power, and functional movements such as the chair sit-to-stand and gait speed. Further, The investigators will evaluate the impact of each protocol on cognitive function.

DETAILED DESCRIPTION:
Resistance training has been shown to have a significant impact on strength, power, cognition, functionality, activities of daily living, and quality of life throughout the aging process(Hunter et al., 2004; Peterson et al., 2010; Wen et al., 2011). Specifically, power training is especially beneficial to older adults to combat the age-related slowing of movement that occurs. and changes in age-related cognitive decline. However, in evaluating these measures and prescribing a power training program, the deficit on either the load or velocity end of the power spectrum unique to these individuals is often overlooked. Therefore, the evaluation of these components coupled with a custom training program to fit their needs on either the load end or velocity end of the spectrum may provide significant benefit to the functionality of older adults. Additionally, sleep quality has been shown to have a significant impact on cognitive performance(Alhola & Polo-Kantola, 2007) and may impact the changes in cognition that The investigators observe with a resistance training program.

Further, muscle mass has been shown to decrease with aging as a result of a variety of physiological changes that occur in the body, including the reduction in motor units and muscle fibers and these changes have a significant impact on the mobility of older adults(Charlier et al., 2016; Evans & Campbell, 1993). Resistance training has been shown to have an impact on the progression and development of sarcopenia and has been supported in the research with both the use of power and strength training programs(Balachandran et al., 2014; Roth et al., 2000). Ultrasonography evaluation of muscle quality can provide valuable information on the changes to the musculature that occur with training programs in older adults(Pardo et al., 2018).

While the impact of power and strength training on muscle quality has been shown(Ivey et al., 2000; Nogueira et al., 2009), the impact of a unique load velocity design to target power deficits on muscle quality is prohibitive. Therefore, this research is designed to evaluate the impact of load training and velocity training on muscle quality in healthy, older adults as well as changes in functionality, cognition, and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Montreal Cognitive Assessment (MOCA) > 23 and no memory loss complaints.

Exclusion Criteria:

* Any uncontrolled cardiovascular or neuromuscular diseases that prevent participation in a training program; Any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, system lupus erythematosus, or other serious concomitant medical illness; Unresolved injury or surgery to the quadricep muscles

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Five-time sit-to-stand | 5 minutes
  The participant will sit with their arms folded across their chest and their back against the chair. On verbal command, the participant will stand up and sit down 5 times as quickly as possible. Timing begins at "Go" and ends when the buttocks touches the chair after the 5th repetition. One practice and two testing trials will be performed.
10-meter walk | 5 minutes
  The participants will be asked to walk as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when they cross the 10-m mark. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed, and the average will be documented in m·s-1. One-minute recoveries will be provided between trials.
One-repetition maximum (1RM) testing | 10 minutes
  One-repetition maximum (1RM) strength testing will include leg press and chest press. After a warm-up, the subject do 10 repetitions a low resistance. The test will begin using a weight near the predicted maximum. The weight will then be increased or decreased depending on the subject's ability to perform the repetition using correct technique.
Home Sleep Testing | 8 hours
  Study participants will have a home sleep study using the NoxA1 system that allows for monitoring of sleep (i.e., EEG) along with respiratory effort and oxygen saturation. The goal of the home sleep study is to exclude other respiratory-related sleep disorders, such as central sleep apnea and Cheyne-Stokes breathing, and efficiently characterize OSA severity. These sleep assessments are routinely done in clinical practice and will be conducted by the participant at home using self-applied portable monitors that are powered by one AA battery. This will only be worn for one night and instruction on setup will be given at the laboratory with a take-home packet for setup.
Actigraphy | 168 hours
  An actigraph, which measures activity levels, will be worn on the wrist for seven consecutive 24-hour periods, to collect data on habitual sleep duration. Wrist actigraphy is a technique for measuring movement over an extended recording period (days to weeks). Data garnered from wrist actigraphy will be used to derive variables such as habitual total sleep time, number and duration of awakenings per night, and napping behavior.

SECONDARY OUTCOMES:
Dimensional Card Sort (DCCS) | 5 minutes
  This is an iPad-administered task (by a research assistant) that measures the flexible use of rules to govern behavior as a means of providing an index of executive function development. The DCCS is a measure of cognitive flexibility. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). "Switch" trials are also employed, in which the participant must change the dimension being matched. For example, after four straight trials the subject is correct on matching shapes, the participant may be asked to match on color on the next trial and then go back to shape, thus requiring the cognitive flexibility to quickly choose the correct stimulus.
Flanker test | 5 minutes
  The Flanker Test uses response inhibition to assess a subject's capacity to suppress incorrect responses within a particular context. The target (in our case an arrow) is flanked by non-target arrows that are either in the same direction as the target (congruent flankers), the opposite response (incongruent flankers), or to neither (neutral flankers).
Picture Sequence Memory Test (PSMT) | 5 minutes
  The PSMT can test episodic memory in persons from 3 through 85. The PSMT involves presentation of sequences of pictured objects and activities in a fixed order on a computer screen and simultaneously verbally described, that the participant must remember and then reproduce over three learning trials.
List Sorting Test | 5 minutes
  The List Sorting Working Memory Test assesses working memory and is part of the NIH Toolbox Cognition Battery. List Sorting is a sequencing task requiring subjects to sort and sequence stimuli that are presented visually and auditorily. Lists may include animal to be sorted by size, foods to be sorted by size, or a combination of the two to be sorted by size.
Pattern Comparison Test | 5 minutes
  The Toolbox Pattern Comparison Processing Speed Test is the assessment of choice to measure reaction time in older adults and is also used to measure processing speed. During the test, participants are asked to identify whether two visual patterns are the "same" or "not the same." Scores reflect the number of correct responses within a finite time frame.
Power Testing | 15 minutes
  Power testing will begin with a warm-up of 10 repetitions at 30% 1RM, followed by a 1-minute recovery period. A second warm-up of 5 repetitions at 30% 1RM will then be performed as rapidly as possible. Peak muscle power will then be assessed at 8 relative intensities (40, 50, 60, 70, and 80% 1RM) on the same resistance machines used for strength testing. The percentages will be randomized to reduce any order effect. For each repetition, the concentric phase will be performed as fast as possible, and the eccentric phase will be performed over 2-3 seconds. Each repetition will be verbally cued "3.2.1. Go!" This testing protocol is commonly used for power testing. Any repetition not performed properly will be repeated after a 1-minute break. Power output will be recorded from the display of each machine and cross-referenced with the electronic spreadsheets. Power testing for leg press and chest press, which are to be used as variables in our analysis, will occur before the beginning
Ultrasound measurement | 15 minutes
  Ultrasound images of the quadriceps femoris muscle (vastus medialis, vastus lateralis, vastus intermedius, rectus femoris) will be taken on the thigh at the two-thirds and midpoint of the length between the anterior superior iliac spine and the upper border of the patella. A LOGIQ P9 R3 Ultrasound System (GE Healthcare, Buckinghamshire, UK) and 3-12 MHz linear array transducer probe will be used, and testing will be conducted on a padded treatment table. Care will be taken to maintain the same standardized body positions and probe locations for all participants. Minimal pressure will be applied by the researcher to reduce any tissue compression that would artificially influence the results. Before acquiring measurements, subjects will rest on the examination table for five minutes to avoid any potential movement-induced stiffness. To improve acoustic contact between the probe and skin, a water-soluble transmission gel will be used on the head of the probe. Both legs will be imaged.
Isokinetic Testing | 30 minutes
  The Biodex 4 Dynamometer will be used for all isokinetic testing. Subjects will be asked to perform an isokinetic warmup of 10 repetitions of leg extension at 270 deg/s, be given a three-minute recovery, and then perform three maximal isokinetic quadriceps extensions at 90, 180, and 300 degrees/second using 2-minute recoveries in between sets. All results will be recorded. The repetitions producing the highest peak torque among the three efforts, and the average power for the repetitions will be used for statistical evaluation. Given the nature of isokinetic testing the resistance is at the speeds we have chosen, far below maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No